CLINICAL TRIAL: NCT00621322
Title: Dose Range Study Evaluating Safety and Immunogenicity Study of GSK Biologicals' Candidate Tuberculosis Vaccines (692342) When Administered to Healthy Adults Aged 18 to 45 Years.
Brief Title: Safety and Immunogenicity Study of GSK Biologicals Tuberculosis Vaccines (692342) to Healthy Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 110345
Record Dates: First submitted 2008-02-12; First posted 2008-02-22 (Estimated); Results first posted 2017-02-03 (Estimated); Last update posted 2018-08-24 (Actual); Status verified 2018-07

CONDITIONS: Tuberculosis
Keywords: Tuberculosis vaccine
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (6):
- Control Group (Placebo Comparator): Healthy adults between and including 18 to 45 years of age at the time of first vaccination, who received 2 doses of the control GSK Biologicals' AS01B adjuvanted system, at Day 0, intramuscularly in the non-dominant arm and at Day 30, intramuscularly in the dominant arm.
  Interventions: Biological: GSK Biologicals' AS01B adjuvant
- GSK692342_F1 Group (Active Comparator): Healthy adults between and including 18 to 45 years of age at the time of first vaccination, who received 2 doses of the non-adjuvanted GSK692342 vaccine formulation 1 (F1), at Day 0, intramuscularly in the non-dominant arm and at Day 30, intramuscularly in the dominant arm.
  Interventions: Biological: GSK Biologicals' Candidate Tuberculosis Vaccine (692342) - Formulation 1
- GSK692342_F2 Group (Experimental): Healthy adults between and including 18 to 45 years of age at the time of first vaccination, who received 2 doses of the adjuvanted GSK692342 vaccine formulation 2 (F2), at Day 0, intramuscularly in the non-dominant arm and at Day 30, intramuscularly in the dominant arm.
  Interventions: Biological: GSK Biologicals' Candidate Tuberculosis Vaccine (692342) - Formulation 2
- GSK692342_F3 Group (Experimental): Healthy adults between and including 18 to 45 years of age at the time of first vaccination, who received 2 doses of the adjuvanted GSK692342 vaccine formulation 3, at Day 0, intramuscularly in the non-dominant arm and at Day 30, intramuscularly in the dominant arm.
  Interventions: Biological: GSK Biologicals' Candidate Tuberculosis Vaccine (692342) - Formulation 3
- GSK692342_F4D1 Group (Experimental): Healthy adults between and including 18 to 45 years of age at the time of first vaccination, who received 2 doses of the adjuvanted GSK692342 vaccine formulation 4 dosage 1 (F4D1), at Day 0, intramuscularly in the non-dominant arm and at Day 30, intramuscularly in the dominant arm.
  Interventions: Biological: GSK Biologicals' Candidate Tuberculosis Vaccine (692342) - Formulation 4 - Dosage 1
- GSK692342_F4D2 Group (Experimental): Healthy adults between and including 18 to 45 years of age at the time of first vaccination, who received 2 doses of the adjuvanted GSK692342 vaccine formulation 4 dosage 2 (F4D2), at Day 0, intramuscularly in the non-dominant arm and at Day 30, intramuscularly in the dominant arm.
  Interventions: Biological: GSK Biologicals' Candidate Tuberculosis Vaccine (692342) - Formulation 4 - Dosage 2

INTERVENTIONS:
Biological: GSK Biologicals' AS01B adjuvant — Intramuscular injection, 2 doses
  Arms: Control Group
Biological: GSK Biologicals' Candidate Tuberculosis Vaccine (692342) - Formulation 1 — Intramuscular injection, 2 doses
  Arms: GSK692342_F1 Group
Biological: GSK Biologicals' Candidate Tuberculosis Vaccine (692342) - Formulation 2 — Intramuscular injection, 2 doses
  Arms: GSK692342_F2 Group
Biological: GSK Biologicals' Candidate Tuberculosis Vaccine (692342) - Formulation 3 — Intramuscular injection, 2 doses
  Arms: GSK692342_F3 Group
Biological: GSK Biologicals' Candidate Tuberculosis Vaccine (692342) - Formulation 4 - Dosage 1 — Intramuscular injection, 2 doses
  Arms: GSK692342_F4D1 Group
Biological: GSK Biologicals' Candidate Tuberculosis Vaccine (692342) - Formulation 4 - Dosage 2 — Intramuscular injection, 2 doses
  Arms: GSK692342_F4D2 Group

SUMMARY:
This observer blind study will assess the safety and immunogenicity of different formulations of GSK Biologicals' 692342 tuberculosis vaccine in healthy adults aged 18 to 45 years with a positive PPD skin test. The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that they can and will comply with the requirements of the protocol should be enrolled in the study.
* A male or female between, and including, 18 and 45 years of age at the time of the first vaccination.
* Written informed consent obtained from the subject prior to any study procedure.
* Free of obvious health problems as established by medical history and clinical examination before enrolment into the study.
* If the subject is female, she must be of non-childbearing potential or if she is of childbearing potential, she must practice adequate contraception for 30 days prior to vaccination, have a negative pregnancy test and continue such precautions for 2 months after completion of the vaccination series.
* No evidence of pulmonary pathology as confirmed by chest X-ray.
* No history of extrapulmonary TB.
* Clinically normal laboratory values for creatinine, alanine aminotransferase (ALT), aspartate aminotransferase (AST), complete blood count (CBC) and urinalysis.
* Seronegative for human immunodeficiency virus-1 and -2 (HIV-1 and -2) antibodies.
* Subjects must have a PPD positive skin reactivity 48 to 72 hours after PPD skin test administration.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose.
* Any chronic drug therapy to be continued during the study period, with the exception of vitamins and/or dietary supplements, herbal medications, birth control pills, anti-histamines for seasonal allergies and SSRIs.
* History of previous administration of experimental Mycobacterium tuberculosis vaccines.
* History of previous exposure to experimental products containing MPL or QS21.
* Administration of any immunoglobulins, any immunotherapy and/or any blood products within the three months preceding the first dose of study vaccination, or planned administrations during the study period.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product (pharmaceutical product or device).
* Any confirmed or suspected immunosuppressive or immunodeficient condition based on medical history and physical examination.
* A family history (first generation) of congenital or hereditary immunodeficiency.
* History of any acute or chronic illness or medication that, in the opinion of the investigator, may interfere with the evaluation of the safety or immunogenicity of the vaccine.
* History of any neurological disorders or seizures.
* History of allergic reactions or anaphylaxis to previous immunisations.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* History of chronic alcohol consumption and/or drug abuse.
* Major congenital defects.
* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2008-04-03 (Actual); Primary Completion 2009-04-03 (Actual); Study Completion 2009-04-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Manila, Philippines

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control Group | GSK692342_F1 Group | GSK692342_F2 Group | GSK692342_F3 Group | GSK692342_F4D1 Group | GSK692342_F4D2 Group
Started | 10 | 10 | 40 | 40 | 40 | 40
Completed | 9 | 10 | 38 | 37 | 39 | 36
Not Completed | 1 | 0 | 2 | 3 | 1 | 4
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 2
Not completed — Migrated/moved from study area | 1 | 0 | 1 | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | GSK692342_F1 Group | GSK692342_F2 Group | GSK692342_F3 Group | GSK692342_F4D1 Group | GSK692342_F4D2 Group | Total
Number analyzed (Participants) | 10 | 10 | 40 | 40 | 40 | 40 | 180
Age, Continuous [Mean (Standard Deviation); unit: Years] | 32.1 (8.10) | 36.0 (5.14) | 30.6 (9.14) | 33.5 (8.73) | 30.6 (9.17) | 31.5 (8.83) | 31.92 (8.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 33 | 36 | 31 | 26 | 142
  Male | 1 | 3 | 7 | 4 | 9 | 14 | 38

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Solicited Local Symptoms
Description: Assessed solicited local symptoms included pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling spreading beyond 50 millimeters (mm) of injection site. Relationship analysis was not performed.
Time Frame: During the 7-day (Days 0-6) post-vaccination period, following each dose and across doses
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects from whom data were available.
Measure: Number; unit: Subjects
Arm/Group | Control Group | GSK692342_F1 Group | GSK692342_F2 Group | GSK692342_F3 Group | GSK692342_F4D1 Group | GSK692342_F4D2 Group
Number analyzed (Participants) | 10 | 10 | 40 | 40 | 40 | 40
Subjects
  Any Pain, Dose 1 | 8 | 3 | 35 | 33 | 33 | 32
  Grade 3 Pain, Dose 1 | 0 | 0 | 0 | 0 | 0 | 1
  Any Redness, Dose 1 | 1 | 2 | 7 | 3 | 4 | 3
  Grade 3 Redness, Dose 1 | 0 | 0 | 0 | 0 | 0 | 0
  Any Swelling, Dose 1 | 0 | 0 | 8 | 6 | 7 | 6
  Grade 3 Swelling, Dose 1 | 0 | 0 | 0 | 0 | 0 | 1
  Any Pain, Dose 2 | 7 | 4 | 33 | 32 | 36 | 33
  Grade 3 Pain, Dose 2 | 0 | 0 | 0 | 0 | 0 | 1
  Any Redness, Dose 2 | 0 | 1 | 0 | 5 | 4 | 5
  Grade 3 Redness, Dose 2 | 0 | 0 | 0 | 0 | 1 | 1
  Any Swelling, Dose 2 | 1 | 1 | 5 | 5 | 7 | 8
  Grade 3 Swelling, Dose 2 | 0 | 0 | 0 | 1 | 1 | 1
  Any Pain, Across | 9 | 5 | 38 | 37 | 37 | 36
  Grade 3 Pain, Across | 0 | 0 | 0 | 0 | 0 | 2
  Any Redness, Across | 1 | 2 | 7 | 6 | 6 | 6
  Grade 3 Redness, Across | 0 | 0 | 0 | 0 | 1 | 1
  Any Swelling, Across | 1 | 1 | 10 | 10 | 12 | 12
  Grade 3 Swelling, Across | 0 | 0 | 0 | 1 | 1 | 2

2. Primary Outcome: Number of Subjects With Solicited General Symptoms
Description: Assessed solicited general symptoms included fatigue, temperature [defined as axillary temperature equal to or above 37.5 degrees Celsius (°C)], gastrointestinal symptoms (gastro) [nausea, vomiting, diarrhoea and/or abdominal pain], headache, malaise and myalgia. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever ≥ 39.0 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: During the 7-day (Days 0-6) post-vaccination period, following each dose and across doses
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Control Group | GSK692342_F1 Group | GSK692342_F2 Group | GSK692342_F3 Group | GSK692342_F4D1 Group | GSK692342_F4D2 Group
Number analyzed (Participants) | 10 | 10 | 40 | 40 | 40 | 40
Subjects
  Any Fatigue, Dose 1 | 1 | 1 | 4 | 5 | 7 | 3
  Grade 3 Fatigue, Dose 1 | 0 | 0 | 0 | 0 | 0 | 0
  Related Fatigue, Dose 1 | 0 | 0 | 1 | 3 | 4 | 2
  Any Gastro, Dose 1 | 2 | 3 | 5 | 3 | 5 | 7
  Grade 3 Gastro, Dose 1 | 0 | 0 | 0 | 0 | 0 | 0
  Related Gastro, Dose 1 | 2 | 0 | 3 | 1 | 1 | 2
  Any Headache, Dose 1 | 4 | 4 | 11 | 16 | 15 | 19
  Grade 3 Headache, Dose 1 | 1 | 1 | 0 | 0 | 0 | 0
  Related Headache, Dose 1 | 2 | 0 | 7 | 8 | 7 | 10
  Any Malaise, Dose 1 | 3 | 3 | 9 | 13 | 10 | 18
  Grade 3 Malaise, Dose 1 | 0 | 0 | 0 | 0 | 0 | 0
  Related Malaise, Dose 1 | 2 | 0 | 7 | 8 | 8 | 16
  Any Myalgia, Dose 1 | 1 | 3 | 14 | 10 | 13 | 14
  Grade 3 Myalgia, Dose 1 | 0 | 0 | 0 | 0 | 0 | 0
  Related Myalgia, Dose 1 | 1 | 1 | 9 | 6 | 11 | 13
  Any Temperature, Dose 1 | 2 | 1 | 3 | 2 | 3 | 9
  Grade 3 Temperature, Dose 1 | 0 | 0 | 0 | 0 | 0 | 2
  Related Temperature, Dose 1 | 1 | 0 | 3 | 1 | 2 | 8
  Any Fatigue, Dose 2 | 1 | 1 | 5 | 6 | 8 | 8
  Grade 3 Fatigue, Dose 2 | 0 | 0 | 0 | 0 | 0 | 0
  Related Fatigue, Dose 2 | 1 | 1 | 4 | 3 | 6 | 7
  Any Gastro, Dose 2 | 1 | 1 | 5 | 7 | 8 | 9
  Grade 3 Gastro, Dose 2 | 0 | 0 | 0 | 0 | 1 | 0
  Related Gastro, Dose 2 | 0 | 0 | 1 | 1 | 7 | 8
  Any Headache, Dose 2 | 5 | 3 | 22 | 20 | 29 | 26
  Grade 3 Headache, Dose 2 | 0 | 0 | 1 | 0 | 1 | 1
  Related Headache, Dose 2 | 1 | 1 | 13 | 8 | 24 | 22
  Any Malaise, Dose 2 | 5 | 1 | 22 | 21 | 21 | 25
  Grade 3 Malaise, Dose 2 | 0 | 0 | 1 | 0 | 0 | 1
  Related Malaise, Dose 2 | 4 | 1 | 21 | 17 | 21 | 24
  Any Myalgia, Dose 2 | 3 | 1 | 18 | 21 | 23 | 28
  Grade 3 Myalgia, Dose 2 | 0 | 0 | 1 | 0 | 2 | 1
  Related Myalgia, Dose 2 | 2 | 1 | 18 | 20 | 23 | 28
  Any Temperature, Dose 2 | 3 | 0 | 15 | 8 | 16 | 27
  Grade 3 Temperature, Dose 2 | 0 | 0 | 2 | 0 | 1 | 3
  Related Temperature, Dose 2 | 2 | 0 | 13 | 7 | 15 | 27
  Any Fatigue, Across | 2 | 1 | 7 | 8 | 13 | 10
  Grade 3 Fatigue, Across | 0 | 0 | 0 | 0 | 0 | 0
  Related Fatigue, Across | 1 | 1 | 4 | 6 | 9 | 8
  Any Gastro, Across | 3 | 3 | 8 | 9 | 11 | 10
  Grade 3 Gastro, Across | 0 | 0 | 0 | 0 | 1 | 0
  Related Gastro, Across | 2 | 0 | 4 | 2 | 8 | 8
  Any Headache, Across | 5 | 6 | 25 | 27 | 30 | 26
  Grade 3 Headache, Across | 1 | 1 | 1 | 0 | 1 | 1
  Related Headache, Across | 3 | 1 | 18 | 15 | 24 | 23
  Any Malaise, Across | 5 | 3 | 23 | 25 | 23 | 26
  Grade 3 Malaise, Across | 0 | 0 | 1 | 0 | 0 | 1
  Related Malaise, Across | 5 | 1 | 22 | 21 | 23 | 26
  Any Myalgia, Across | 3 | 3 | 25 | 23 | 24 | 29
  Grade 3 Myalgia, Across | 0 | 0 | 1 | 0 | 2 | 1
  Related Myalgia, Across | 2 | 2 | 24 | 22 | 24 | 29
  Any Temperature, Across | 5 | 1 | 17 | 9 | 17 | 28
  Grade 3 Temperature, Across | 0 | 0 | 2 | 0 | 1 | 4
  Related Temperature, Across | 3 | 0 | 15 | 7 | 15 | 28

3. Primary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Grade 3 AE = an AE which prevented normal, everyday activities. Related = AE assessed by the investigator as related to the vaccination.
Time Frame: During the 30-day (Days 0-29) post-vaccination period
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Control Group | GSK692342_F1 Group | GSK692342_F2 Group | GSK692342_F3 Group | GSK692342_F4D1 Group | GSK692342_F4D2 Group
Number analyzed (Participants) | 10 | 10 | 40 | 40 | 40 | 40
Subjects
  Any AEs | 7 | 9 | 29 | 33 | 33 | 27
  Grade 3 AEs | 0 | 0 | 1 | 1 | 0 | 0
  Related AEs | 0 | 1 | 7 | 2 | 5 | 2

4. Primary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: During the entire study period (from Day 0 up to Day 210)
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Control Group | GSK692342_F1 Group | GSK692342_F2 Group | GSK692342_F3 Group | GSK692342_F4D1 Group | GSK692342_F4D2 Group
Number analyzed (Participants) | 10 | 10 | 40 | 40 | 40 | 40
Subjects | 0 | 0 | 2 | 0 | 2 | 0

5. Primary Outcome: Number of Subjects With Different Biochemical and Haematological Levels
Description: Among biochemical and haematological parameters assessed were alanine aminotransferase [ALT], aspartate aminotransferase [AST], basophils [BAS], creatinine [CREA], eosinophils [EOS], haematocrit [Hct], haemoglobin [Hgb], lymphocytes [LYM], monocytes [MON], neutrophils [NEU], platelets [PLA], red blood cells [RBC] and white blood cells [WBC]. Levels of haematological/biochemical parameters assessed in terms of normal laboratory values were- normal, below and above.
Time Frame: At Day 0
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Control Group | GSK692342_F1 Group | GSK692342_F2 Group | GSK692342_F3 Group | GSK692342_F4D1 Group | GSK692342_F4D2 Group
Number analyzed (Participants) | 10 | 10 | 40 | 40 | 40 | 40
Subjects
  ALT, Normal | 10 | 10 | 40 | 38 | 38 | 37
  ALT, Below | 0 | 0 | 0 | 0 | 0 | 0
  ALT, Above | 0 | 0 | 0 | 1 | 2 | 3
  ALT, Missing | 0 | 0 | 0 | 1 | 0 | 0
  AST, Normal | 9 | 9 | 40 | 38 | 37 | 38
  AST, Below | 0 | 0 | 0 | 0 | 0 | 0
  AST, Above | 1 | 1 | 0 | 1 | 3 | 2
  AST, Missing | 0 | 0 | 0 | 1 | 0 | 0
  BAS, Normal | 3 | 10 | 11 | 18 | 40 | 39
  BAS, Below | 0 | 0 | 0 | 0 | 0 | 0
  BAS, Above | 0 | 0 | 0 | 0 | 0 | 0
  BAS, Missing | 7 | 0 | 29 | 22 | 0 | 1
  CREA, Normal | 9 | 10 | 38 | 38 | 39 | 39
  CREA, Below | 1 | 0 | 2 | 1 | 1 | 1
  CREA, Above | 0 | 0 | 0 | 0 | 0 | 0
  CREA, Missing | 0 | 0 | 0 | 1 | 0 | 0
  EOS, Normal | 9 | 8 | 38 | 38 | 33 | 34
  EOS, Below | 0 | 0 | 1 | 1 | 0 | 0
  EOS, Above | 1 | 2 | 0 | 1 | 7 | 5
  EOS, Missing | 0 | 0 | 1 | 0 | 0 | 1
  Hct, Normal | 10 | 9 | 38 | 39 | 37 | 35
  Hct, Below | 0 | 1 | 1 | 1 | 3 | 4
  Hct, Above | 0 | 0 | 0 | 0 | 0 | 0
  Hct, Missing | 0 | 0 | 1 | 0 | 0 | 1
  Hgb, Normal | 10 | 8 | 39 | 39 | 38 | 36
  Hgb, Below | 0 | 2 | 0 | 1 | 2 | 3
  Hgb, Above | 0 | 0 | 0 | 0 | 0 | 0
  Hgb, Missing | 0 | 0 | 1 | 0 | 0 | 1
  LYM, Normal | 9 | 10 | 38 | 37 | 39 | 37
  LYM, Below | 1 | 0 | 1 | 3 | 1 | 2
  LYM, Above | 0 | 0 | 0 | 0 | 0 | 0
  LYM, Missing | 0 | 0 | 1 | 0 | 0 | 1
  MON, Normal | 10 | 9 | 39 | 40 | 38 | 38
  MON, Below | 0 | 1 | 0 | 0 | 2 | 1
  MON, Above | 0 | 0 | 0 | 0 | 0 | 0
  MON, Missing | 0 | 0 | 1 | 0 | 0 | 1
  NEU, Normal | 9 | 10 | 35 | 36 | 37 | 36
  NEU, Below | 0 | 0 | 0 | 0 | 0 | 0
  NEU, Above | 1 | 0 | 4 | 4 | 3 | 3
  NEU, Missing | 0 | 0 | 1 | 0 | 0 | 1
  PLA, Normal | 10 | 10 | 39 | 40 | 40 | 39
  PLA, Below | 0 | 0 | 0 | 0 | 0 | 0
  PLA, Above | 0 | 0 | 0 | 0 | 0 | 0
  PLA, Missing | 0 | 0 | 1 | 0 | 0 | 1
  RBC, Normal | 9 | 7 | 36 | 35 | 36 | 35
  RBC, Below | 1 | 1 | 2 | 1 | 2 | 4
  RBC, Above | 0 | 2 | 1 | 4 | 2 | 0
  RBC, Missing | 0 | 0 | 1 | 0 | 0 | 1
  WBC, Normal | 10 | 9 | 37 | 31 | 30 | 36
  WBC, Below | 0 | 0 | 0 | 0 | 1 | 0
  WBC, Above | 0 | 1 | 2 | 9 | 9 | 3
  WBC, Missing | 0 | 0 | 1 | 0 | 0 | 1

6. Primary Outcome: Number of Subjects With Different Biochemical and Haematological Levels
Description: as for outcome 5
Time Frame: At Day 7
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Control Group | GSK692342_F1 Group | GSK692342_F2 Group | GSK692342_F3 Group | GSK692342_F4D1 Group | GSK692342_F4D2 Group
Number analyzed (Participants) | 10 | 10 | 40 | 40 | 40 | 40
Subjects
  ALT, Normal | 10 | 10 | 36 | 32 | 38 | 34
  ALT, Below | 0 | 0 | 1 | 0 | 0 | 1
  ALT, Above | 0 | 0 | 2 | 7 | 2 | 4
  ALT, Missing | 0 | 0 | 0 | 1 | 0 | 0
  AST, Normal | 10 | 10 | 39 | 36 | 40 | 37
  AST, Below | 0 | 0 | 0 | 0 | 0 | 0
  AST, Above | 0 | 0 | 0 | 3 | 0 | 2
  AST, Missing | 0 | 0 | 1 | 1 | 1 | 1
  BAS, Normal | 2 | 10 | 1 | 7 | 40 | 39
  BAS, Below | 0 | 0 | 0 | 0 | 0 | 0
  BAS, Above | 0 | 0 | 0 | 0 | 0 | 0
  BAS, Missing | 8 | 0 | 39 | 33 | 0 | 1
  CREA, Normal | 10 | 10 | 38 | 36 | 39 | 39
  CREA, Below | 0 | 0 | 0 | 0 | 1 | 0
  CREA, Above | 0 | 0 | 1 | 3 | 0 | 0
  CREA, Missing | 0 | 0 | 1 | 1 | 0 | 1
  EOS, Normal | 10 | 6 | 38 | 38 | 32 | 31
  EOS, Below | 0 | 0 | 0 | 0 | 0 | 0
  EOS, Above | 0 | 4 | 1 | 2 | 8 | 8
  EOS, Missing | 0 | 0 | 1 | 0 | 0 | 1
  Hct, Normal | 10 | 8 | 37 | 37 | 34 | 33
  Hct, Below | 0 | 2 | 2 | 3 | 6 | 6
  Hct, Above | 0 | 0 | 0 | 0 | 0 | 0
  Hct, Missing | 0 | 0 | 1 | 0 | 0 | 1
  Hgb, Normal | 10 | 7 | 39 | 38 | 33 | 36
  Hgb, Below | 0 | 3 | 0 | 2 | 7 | 3
  Hgb, Above | 0 | 0 | 0 | 0 | 0 | 0
  Hgb, Missing | 0 | 0 | 1 | 0 | 0 | 1
  LYM, Normal | 10 | 10 | 38 | 40 | 40 | 38
  LYM, Below | 0 | 0 | 1 | 0 | 0 | 1
  LYM, Above | 0 | 0 | 0 | 0 | 0 | 0
  LYM, Missing | 0 | 0 | 1 | 0 | 0 | 1
  MON, Normal | 10 | 9 | 39 | 40 | 38 | 39
  MON, Below | 0 | 1 | 0 | 0 | 2 | 0
  MON, Above | 0 | 0 | 0 | 0 | 0 | 0
  MON, Missing | 0 | 0 | 1 | 0 | 0 | 1
  NEU, Normal | 9 | 10 | 38 | 40 | 40 | 38
  NEU, Below | 0 | 0 | 0 | 0 | 0 | 0
  NEU, Above | 1 | 0 | 1 | 0 | 0 | 1
  NEU, Missing | 0 | 0 | 1 | 0 | 0 | 1
  PLA, Normal | 10 | 9 | 39 | 40 | 39 | 39
  PLA, Below | 0 | 0 | 0 | 0 | 0 | 0
  PLA, Above | 0 | 1 | 0 | 0 | 1 | 0
  PLA, Missing | 0 | 0 | 1 | 0 | 0 | 1
  RBC, Normal | 8 | 8 | 33 | 33 | 34 | 33
  RBC, Below | 2 | 1 | 5 | 5 | 5 | 6
  RBC, Above | 0 | 1 | 1 | 2 | 1 | 0
  RBC, Missing | 0 | 0 | 1 | 0 | 0 | 1
  WBC, Normal | 9 | 9 | 33 | 37 | 31 | 35
  WBC, Below | 0 | 0 | 0 | 0 | 2 | 0
  WBC, Above | 1 | 1 | 6 | 3 | 7 | 4
  WBC, Missing | 0 | 0 | 1 | 0 | 0 | 1

7. Primary Outcome: Number of Subjects With Different Biochemical and Haematological Levels
Description: as for outcome 5
Time Frame: At Day 30
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Control Group | GSK692342_F1 Group | GSK692342_F2 Group | GSK692342_F3 Group | GSK692342_F4D1 Group | GSK692342_F4D2 Group
Number analyzed (Participants) | 10 | 10 | 40 | 40 | 40 | 40
Subjects
  ALT, Normal | 9 | 9 | 38 | 36 | 36 | 38
  ALT, Below | 0 | 0 | 0 | 0 | 1 | 0
  ALT, Above | 1 | 1 | 1 | 2 | 3 | 1
  ALT, Missing | 0 | 0 | 1 | 2 | 0 | 1
  AST, Normal | 10 | 10 | 38 | 35 | 37 | 37
  AST, Below | 0 | 0 | 0 | 0 | 0 | 0
  AST, Above | 0 | 0 | 1 | 3 | 3 | 2
  AST, Missing | 0 | 0 | 1 | 2 | 0 | 1
  BAS, Normal | 4 | 10 | 5 | 13 | 39 | 39
  BAS, Below | 0 | 0 | 0 | 0 | 0 | 0
  BAS, Above | 0 | 0 | 0 | 0 | 0 | 0
  BAS, Missing | 6 | 0 | 35 | 27 | 1 | 1
  CREA, Normal | 10 | 9 | 39 | 37 | 36 | 37
  CREA, Below | 0 | 0 | 0 | 0 | 3 | 0
  CREA, Above | 0 | 1 | 0 | 1 | 1 | 2
  CREA, Missing | 0 | 0 | 1 | 2 | 0 | 1
  EOS, Normal | 8 | 8 | 37 | 35 | 28 | 30
  EOS, Below | 0 | 0 | 1 | 0 | 0 | 0
  EOS, Above | 1 | 2 | 1 | 5 | 11 | 9
  EOS, Missing | 1 | 0 | 1 | 0 | 1 | 1
  Hct, Normal | 8 | 7 | 36 | 34 | 34 | 35
  Hct, Below | 1 | 3 | 3 | 5 | 5 | 4
  Hct, Above | 0 | 0 | 0 | 1 | 0 | 0
  Hct, Missing | 1 | 0 | 1 | 0 | 1 | 1
  Hgb, Normal | 8 | 7 | 38 | 35 | 33 | 36
  Hgb, Below | 1 | 3 | 1 | 4 | 6 | 3
  Hgb, Above | 0 | 0 | 0 | 1 | 0 | 0
  Hgb, Missing | 1 | 0 | 1 | 0 | 1 | 1
  LYM, Normal | 9 | 9 | 38 | 40 | 39 | 36
  LYM, Below | 0 | 1 | 1 | 0 | 0 | 3
  LYM, Above | 0 | 0 | 0 | 0 | 0 | 0
  LYM, Missing | 1 | 0 | 1 | 0 | 1 | 1
  MON, Normal | 9 | 10 | 39 | 40 | 39 | 39
  MON, Below | 0 | 0 | 0 | 0 | 0 | 0
  MON, Above | 0 | 0 | 0 | 0 | 0 | 0
  MON, Missing | 1 | 0 | 1 | 0 | 1 | 1
  NEU, Normal | 9 | 10 | 38 | 39 | 38 | 39
  NEU, Below | 0 | 0 | 0 | 0 | 0 | 0
  NEU, Above | 0 | 0 | 1 | 1 | 1 | 0
  NEU, Missing | 1 | 0 | 1 | 0 | 1 | 1
  PLA, Normal | 9 | 10 | 39 | 40 | 38 | 39
  PLA, Below | 0 | 0 | 0 | 0 | 1 | 0
  PLA, Above | 0 | 0 | 0 | 0 | 0 | 0
  PLA, Missing | 1 | 0 | 1 | 0 | 1 | 1
  RBC, Normal | 9 | 8 | 36 | 36 | 36 | 36
  RBC, Below | 0 | 1 | 2 | 2 | 2 | 3
  RBC, Above | 0 | 1 | 1 | 2 | 1 | 0
  RBC, Missing | 1 | 0 | 1 | 0 | 1 | 1
  WBC, Normal | 9 | 8 | 35 | 37 | 33 | 36
  WBC, Below | 0 | 0 | 0 | 0 | 3 | 0
  WBC, Above | 0 | 2 | 4 | 3 | 3 | 3
  WBC, Missing | 1 | 0 | 1 | 0 | 1 | 1

8. Primary Outcome: Number of Subjects With Different Biochemical and Haematological Levels
Description: as for outcome 5
Time Frame: At Day 37
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Control Group | GSK692342_F1 Group | GSK692342_F2 Group | GSK692342_F3 Group | GSK692342_F4D1 Group | GSK692342_F4D2 Group
Number analyzed (Participants) | 10 | 10 | 40 | 40 | 40 | 40
Subjects
  ALT, Normal | 9 | 10 | 37 | 36 | 34 | 35
  ALT, Below | 0 | 0 | 0 | 0 | 0 | 0
  ALT, Above | 1 | 0 | 2 | 3 | 6 | 4
  ALT, Missing | 0 | 0 | 1 | 1 | 0 | 1
  AST, Normal | 10 | 10 | 37 | 38 | 37 | 36
  AST, Below | 0 | 0 | 0 | 0 | 0 | 0
  AST, Above | 0 | 0 | 2 | 1 | 3 | 3
  AST, Missing | 0 | 0 | 1 | 1 | 1 | 1
  BAS, Normal | 4 | 10 | 10 | 15 | 40 | 39
  BAS, Below | 0 | 0 | 0 | 0 | 0 | 0
  BAS, Above | 0 | 0 | 0 | 0 | 0 | 0
  BAS, Missing | 6 | 0 | 0 | 25 | 0 | 1
  CREA, Normal | 10 | 9 | 38 | 39 | 38 | 39
  CREA, Above | 0 | 0 | 0 | 0 | 2 | 0
  CREA, Below | 0 | 1 | 1 | 0 | 0 | 0
  CREA, Missing | 0 | 0 | 1 | 1 | 0 | 1
  EOS, Normal | 6 | 7 | 35 | 36 | 33 | 33
  EOS, Below | 0 | 0 | 1 | 0 | 0 | 0
  EOS, Above | 4 | 3 | 3 | 3 | 7 | 6
  EOS, Missing | 0 | 0 | 1 | 1 | 0 | 1
  Hct, Normal | 8 | 7 | 34 | 32 | 35 | 35
  Hct, Below | 2 | 3 | 5 | 6 | 5 | 4
  Hct, Above | 0 | 0 | 0 | 1 | 0 | 0
  Hct, Missing | 0 | 0 | 1 | 1 | 0 | 1
  Hgb, Normal | 9 | 6 | 36 | 34 | 36 | 36
  Hgb, Below | 1 | 4 | 3 | 4 | 4 | 3
  Hgb, Above | 0 | 0 | 0 | 1 | 0 | 0
  Hgb, Missing | 0 | 0 | 1 | 1 | 0 | 1
  LYM, Normal | 10 | 10 | 38 | 38 | 39 | 39
  LYM, Below | 0 | 0 | 1 | 0 | 1 | 0
  LYM, Above | 0 | 0 | 0 | 1 | 0 | 0
  LYM, Missing | 0 | 0 | 1 | 1 | 0 | 1
  MON, Normal | 10 | 10 | 39 | 38 | 39 | 39
  MON, Below | 0 | 0 | 0 | 0 | 1 | 0
  MON, Above | 0 | 0 | 0 | 1 | 0 | 0
  MON, Missing | 0 | 0 | 1 | 1 | 0 | 1
  NEU, Normal | 10 | 10 | 38 | 38 | 39 | 37
  NEU, Below | 0 | 0 | 0 | 1 | 0 | 1
  NEU, Above | 0 | 0 | 1 | 0 | 1 | 1
  NEU, Missing | 0 | 0 | 1 | 1 | 0 | 1
  PLA, Normal | 10 | 9 | 37 | 39 | 40 | 39
  PLA, Below | 0 | 0 | 0 | 0 | 0 | 0
  PLA, Above | 0 | 1 | 2 | 0 | 0 | 0
  PLA, Missing | 0 | 0 | 1 | 1 | 0 | 1
  RBC, Normal | 9 | 8 | 34 | 35 | 36 | 33
  RBC, Below | 1 | 1 | 5 | 2 | 3 | 6
  RBC, Above | 0 | 1 | 0 | 2 | 1 | 0
  RBC, Missing | 0 | 0 | 1 | 1 | 0 | 1
  WBC, Normal | 9 | 7 | 32 | 35 | 33 | 34
  WBC, Below | 0 | 0 | 0 | 1 | 0 | 0
  WBC, Above | 1 | 3 | 7 | 3 | 7 | 5
  WBC, Missing | 0 | 0 | 1 | 1 | 0 | 1

9. Primary Outcome: Number of Subjects With Different Biochemical and Haematological Levels
Description: as for outcome 5
Time Frame: At Day 60
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Control Group | GSK692342_F1 Group | GSK692342_F2 Group | GSK692342_F3 Group | GSK692342_F4D1 Group | GSK692342_F4D2 Group
Number analyzed (Participants) | 10 | 10 | 40 | 40 | 40 | 40
Subjects
  ALT, Normal | 9 | 9 | 38 | 37 | 38 | 34
  ALT, Below | 0 | 0 | 0 | 0 | 0 | 0
  ALT, Above | 1 | 1 | 1 | 2 | 2 | 5
  ALT, Missing | 0 | 0 | 1 | 1 | 0 | 1
  AST, Normal | 9 | 9 | 38 | 37 | 38 | 37
  AST, Below | 0 | 0 | 0 | 0 | 0 | 0
  AST, Above | 1 | 1 | 1 | 2 | 2 | 2
  AST, Missing | 0 | 0 | 1 | 1 | 0 | 1
  BAS, Normal | 10 | 10 | 38 | 39 | 40 | 39
  BAS, Below | 0 | 0 | 0 | 0 | 0 | 0
  BAS, Above | 0 | 0 | 0 | 0 | 0 | 0
  BAS, Missing | 0 | 0 | 2 | 1 | 0 | 1
  CREA, Normal | 10 | 9 | 38 | 37 | 39 | 39
  CREA, Below | 0 | 1 | 1 | 2 | 1 | 0
  CREA, Above | 0 | 0 | 0 | 0 | 0 | 0
  CREA, Missing | 0 | 0 | 1 | 1 | 0 | 1
  EOS, Normal | 7 | 7 | 34 | 36 | 32 | 31
  EOS, Below | 0 | 0 | 0 | 0 | 0 | 0
  EOS, Above | 3 | 3 | 4 | 3 | 8 | 8
  EOS, Missing | 0 | 0 | 2 | 1 | 0 | 1
  Hct, Normal | 9 | 8 | 33 | 36 | 36 | 36
  Hct, Below | 1 | 2 | 5 | 2 | 4 | 3
  Hct, Above | 0 | 0 | 0 | 1 | 0 | 0
  Hct, Missing | 0 | 0 | 2 | 1 | 0 | 1
  Hgb, Normal | 9 | 8 | 35 | 36 | 37 | 36
  Hgb, Below | 1 | 2 | 3 | 2 | 3 | 3
  Hgb, Above | 0 | 0 | 0 | 1 | 0 | 0
  Hgb, Missing | 0 | 0 | 2 | 1 | 0 | 1
  LYM, Normal | 10 | 8 | 38 | 39 | 38 | 37
  LYM, Below | 0 | 2 | 0 | 0 | 2 | 2
  LYM, Above | 0 | 0 | 0 | 0 | 0 | 0
  LYM, Missing | 0 | 0 | 2 | 1 | 0 | 1
  MON, Normal | 10 | 9 | 37 | 39 | 40 | 39
  MON, Below | 0 | 1 | 1 | 0 | 0 | 0
  MON, Above | 0 | 0 | 0 | 0 | 0 | 0
  MON, Missing | 0 | 0 | 2 | 1 | 0 | 1
  NEU, Normal | 9 | 8 | 38 | 39 | 37 | 37
  NEU, Below | 0 | 0 | 0 | 0 | 0 | 0
  NEU, Above | 1 | 2 | 0 | 0 | 3 | 2
  NEU, Missing | 0 | 0 | 2 | 1 | 0 | 1
  PLA, Normal | 10 | 9 | 38 | 38 | 40 | 39
  PLA, Below | 0 | 0 | 0 | 0 | 0 | 0
  PLA, Above | 0 | 1 | 0 | 1 | 0 | 0
  PLA, Missing | 0 | 0 | 2 | 1 | 0 | 1
  RBC, Normal | 9 | 8 | 36 | 35 | 37 | 36
  RBC, Below | 1 | 1 | 2 | 3 | 2 | 3
  RBC, Above | 0 | 1 | 0 | 1 | 1 | 0
  RBC, Missing | 0 | 0 | 2 | 1 | 0 | 1
  WBC, Normal | 8 | 7 | 34 | 37 | 36 | 31
  WBC, Below | 0 | 0 | 0 | 0 | 1 | 1
  WBC, Above | 2 | 3 | 4 | 2 | 3 | 7
  WBC, Missing | 0 | 0 | 2 | 1 | 0 | 1

10. Secondary Outcome: Frequency of Mycobacterium Tuberculosis Fusion Protein (M72) Specific Cluster of Differentiation 4/8 (CD4/8+) T Cells Expressing at Least Two Different Cytokines
Description: Among cytokines expressed were interleukin-2 [IL-2] and/or interferon-gamma [IFN-γ] and/or tumour necrosis factor-alpha [TNF-α] and/or cluster of differentiation 40-ligand [CD40-L]. Analysis of cytokines expression was done by means of in vitro flow cytometry, using intracellular cytokine staining (ICS).
Time Frame: At Day 0, 30, 60 and 210
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects for whom data concerning immunogenicity outcome variables were available.
Measure: Median (Inter-Quartile Range); unit: T cells/million cells
Arm/Group | Control Group | GSK692342_F1 Group | GSK692342_F2 Group | GSK692342_F3 Group | GSK692342_F4D1 Group | GSK692342_F4D2 Group
Number analyzed (Participants) | 10 | 10 | 40 | 40 | 40 | 40
T cells/million cells
  CD4-All Doubles, D0 [N=9;9;38;34;40;39] | 173.0 [94.0 to 466.0] | 293.0 [213.0 to 853.0] | 200.0 [87.0 to 537.0] | 241.0 [147.0 to 547.0] | 263.5 [80.5 to 528.5] | 312.0 [133.0 to 488.0]
  CD4-All Doubles, D30 [N=10;10;38;36;39;37] | 245.5 [80.0 to 387.0] | 1013.5 [491.0 to 3227.0] | 2833.0 [1440.0 to 5120.0] | 1653.5 [886.5 to 3587.0] | 2653.0 [1480.0 to 4826.0] | 3280.0 [2267.0 to 6928.0]
  CD4-All Doubles, D60 [N=10;9;38;36;38;37] | 139.5 [27.0 to 187.0] | 2133.0 [640.0 to 3240.0] | 6307.0 [3560.0 to 9307.0] | 3855.5 [2353.5 to 5220.0] | 4880.0 [3147.0 to 6853.0] | 5133.0 [3227.0 to 7733.0]
  CD4-All Doubles, D210 [N=9;7;37;32;35;34] | 106.0 [91.0 to 414.0] | 1426.0 [949.0 to 2814.0] | 3826.0 [2467.0 to 5907.0] | 2486.5 [1660.0 to 4075.0] | 3240.0 [2520.0 to 5360.0] | 3633.5 [2733.0 to 5253.0]
  CD8-All Doubles, D0 [N=9;9;38;34;40;39] | 1.0 [1.0 to 65.0] | 5.0 [1.0 to 35.0] | 17.0 [1.0 to 104.0] | 33.0 [1.0 to 85.0] | 9.0 [1.0 to 91.0] | 18.0 [1.0 to 79.0]
  CD8-All Doubles, D30 [N=10;10;38;36;39;37] | 31.0 [1.0 to 46.0] | 20.5 [1.0 to 146.0] | 39.5 [1.0 to 102.0] | 14.0 [1.0 to 77.5] | 26.0 [1.0 to 287.0] | 34.0 [1.0 to 90.0]
  CD8-All Doubles, D60 [N=10;9;38;36;38;37] | 9.5 [1.0 to 175.0] | 16.0 [1.0 to 33.0] | 1.0 [1.0 to 71.0] | 10.0 [1.0 to 86.5] | 59.0 [1.0 to 167.0] | 16.0 [1.0 to 107.0]
  CD8-All Doubles, D210 [N=9;7;37;32;35;34] | 1.0 [1.0 to 179.0] | 1.0 [1.0 to 28.0] | 1.0 [1.0 to 35.0] | 1.0 [1.0 to 84.0] | 54.0 [2.0 to 124.0] | 24.5 [1.0 to 46.0]

11. Secondary Outcome: Frequency of M72 Specific CD4/8+ T Cells Expressing at Least One Cytokine and Another Signal Molecule
Description: Expressed cytokine combinations for CD4+ T cells were CD40-L and IL-2 or IFN-γ or TNF-α; IL-2 and CD40-L, or IFN-γ, or TNF-α; IFN-γ and CD40-L, or IL-2, or TNF-α; TNF-α and CD40-L, or IL-2, or IFN-γ.
  For CD8+ T cells no vaccine induced responses were observed, thus results are presented only for the frequency of M72-specific CD8+ T cells expressing at least two cytokines.
Time Frame: At Day 0, 30, 60 and 210
Population: The analysis was performed on the ATP cohort for immunogenicity, which included all evaluable subjects for whom data concerning immunogenicity outcome variables were available.
Measure: Median (Inter-Quartile Range); unit: T cells/million cells
Arm/Group | Control Group | GSK692342_F1 Group | GSK692342_F2 Group | GSK692342_F3 Group | GSK692342_F4D1 Group | GSK692342_F4D2 Group
Number analyzed (Participants) | 10 | 10 | 40 | 40 | 40 | 40
T cells/million cells
  CD4-CD40-L, D0 [N=9;9;38;34;40;39] | 104.0 [66.0 to 306.0] | 227.0 [186.0 to 840.0] | 147.0 [41.0 to 254.0] | 151.0 [107.0 to 320.0] | 210.5 [73.0 to 388.0] | 261.0 [94.0 to 418.0]
  CD4-CD40-L, D30 [N=10;10;38;36;39;37] | 188.0 [40.0 to 307.0] | 853.0 [427.0 to 3133.0] | 1934.0 [1333.0 to 3600.0] | 1280.0 [833.5 to 2219.5] | 2334.0 [1387.0 to 3700.0] | 3213.0 [1853.0 to 6801.0]
  CD4-CD40-L, D60 [N=10;9;38;36;38;37] | 87.0 [1.0 to 227.0] | 1986.0 [560.0 to 3173.0] | 5413.5 [2535.0 to 7235.0] | 2813.5 [1740.0 to 4293.5] | 4384.5 [2826.0 to 5813.0] | 4680.0 [3120.0 to 6547.0]
  CD4-CD40-L, D210 [N=9;7;37;32;35;34] | 120.0 [80.0 to 380.0] | 1374.0 [920.0 to 2693.0] | 3727.0 [2431.0 to 5733.0] | 2424.5 [1586.5 to 3744.0] | 3173.0 [2333.0 to 5307.0] | 3540.0 [2486.0 to 5025.0]
  CD40-IL-2, D0 [N=9;9;38;34;40;39] | 146.0 [93.0 to 467.0] | 333.0 [207.0 to 787.0] | 173.0 [66.0 to 373.0] | 224.0 [80.0 to 477.0] | 202.5 [73.5 to 413.0] | 226.0 [67.0 to 360.0]
  CD4-IL-2, D30 [N=10;10;38;36;39;37] | 218.5 [40.0 to 320.0] | 1046.5 [453.0 to 2356.0] | 2560.0 [1426.0 to 4680.0] | 1460.0 [827.0 to 3093.5] | 2520.0 [1147.0 to 4186.0] | 3120.0 [1806.0 to 6546.0]
  CD4-IL-2, D60 [N=10;9;38;36;38;37] | 107.0 [34.0 to 200.0] | 1773.0 [533.0 to 2840.0] | 5704.0 [3284.0 to 7947.0] | 3068.5 [2055.5 to 4473.0] | 4460.0 [2762.0 to 5591.0] | 4414.0 [2894.0 to 7027.0]
  CD4-IL-2, D210 [N=9;7;37;32;35;34] | 114.0 [66.0 to 312.0] | 1427.0 [840.0 to 2227.0] | 3240.0 [2360.0 to 5813.0] | 2180.0 [1526.5 to 3569.5] | 3080.0 [2293.0 to 5226.0] | 3533.5 [2400.0 to 5037.0]
  CD40-TNF-α, D0 [N=9;9;38;34;40;39] | 78.0 [53.0 to 334.0] | 220.0 [146.0 to 640.0] | 143.5 [67.0 to 493.0] | 180.5 [79.0 to 449.0] | 177.5 [56.0 to 398.0] | 160.0 [29.0 to 293.0]
  CD4-TNF-α, D30 [N=10;10;38;36;39;37] | 185.5 [93.0 to 346.0] | 733.5 [345.0 to 2360.0] | 2028.0 [1013.0 to 4080.0] | 1140.0 [473.5 to 3026.5] | 1534.0 [867.0 to 3813.0] | 2133.0 [867.0 to 4480.0]
  CD4-TNF-α, D60 [N=10;9;38;36;38;37] | 73.0 [1.0 to 226.0] | 907.0 [427.0 to 1373.0] | 3993.5 [1788.0 to 7223.0] | 2086.5 [1306.5 to 3754.0] | 3019.5 [1790.0 to 3776.0] | 2867.0 [1510.0 to 4200.0]
  CD4-TNF-α, D210 [N=9;7;37;32;35;34] | 72.0 [1.0 to 379.0] | 1106.0 [718.0 to 2307.0] | 2960.0 [1613.0 to 4987.0] | 1831.0 [1086.0 to 3096.0] | 2305.0 [1694.0 to 4133.0] | 2580.0 [1840.0 to 4240.0]
  CD40-IFN-γ, D0 [N=9;9;38;34;40;39] | 134.0 [13.0 to 480.0] | 258.0 [214.0 to 840.0] | 180.5 [67.0 to 471.0] | 193.5 [69.0 to 435.0] | 233.5 [67.0 to 493.5] | 306.0 [146.0 to 483.0]
  CD4-IFN-γ, D30 [N=10;10;38;36;39;37] | 206.5 [54.0 to 279.0] | 626.5 [333.0 to 2306.0] | 1477.0 [496.0 to 3675.0] | 938.5 [347.5 to 2500.0] | 1097.0 [654.0 to 3440.0] | 1733.0 [698.0 to 4688.0]
  CD4-IFN-γ, D60 [N=10;9;38;36;38;37] | 111.0 [40.0 to 266.0] | 1014.0 [320.0 to 1480.0] | 3070.5 [1134.0 to 4794.0] | 1233.0 [667.0 to 2946.5] | 2016.0 [1253.0 to 3010.0] | 2453.0 [1320.0 to 3853.0]
  CD4-IFN-γ, D210 [N=9;7;37;32;35;34] | 146.0 [107.0 to 360.0] | 933.0 [336.0 to 1826.0] | 1907.0 [827.0 to 3413.0] | 927.0 [483.5 to 1823.5] | 1413.0 [915.0 to 2054.0] | 1711.0 [892.0 to 2310.0]

12. Secondary Outcome: Anti-M72 Specific Antibody Concentrations
Description: Concentrations given in enzyme-linked immunosorbent assay units per milliliter (EL.U/mL) were expressed as geometric mean concentrations (GMCs).
Time Frame: At Day 0, 30, 60 and 210
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Control Group | GSK692342_F1 Group | GSK692342_F2 Group | GSK692342_F3 Group | GSK692342_F4D1 Group | GSK692342_F4D2 Group
Number analyzed (Participants) | 10 | 10 | 40 | 40 | 40 | 40
EL.U/mL
  Anti-M72, D0 [N=10;10;39;38;40;39] | 1.4 [1.4 to 1.4] | 1.4 [1.4 to 1.4] | 1.4 [1.4 to 1.4] | 1.4 [1.4 to 1.4] | 1.4 [1.4 to 1.4] | 1.4 [1.4 to 1.4]
  Anti-M72, D30 [N=10;10;39;38;40;39] | 1.4 [1.4 to 1.4] | 2.9 [1.4 to 6.0] | 4.9 [3.5 to 6.9] | 5.5 [4.1 to 7.4] | 8.7 [6.5 to 11.7] | 15.0 [11.2 to 20.0]
  Anti-M72, D60 [N=10;10;39;38;40;39] | 1.4 [1.4 to 1.4] | 31.0 [7.3 to 132.0] | 458.4 [365.2 to 575.4] | 468.5 [367.0 to 598.0] | 598.6 [504.0 to 710.9] | 833.0 [696.2 to 996.7]
  Anti-M72, D210 [N=9;10;38;36;39;36] | 1.4 [1.4 to 1.4] | 6.1 [2.1 to 17.8] | 51.1 [37.5 to 69.8] | 46.3 [37.2 to 57.6] | 70.7 [57.5 to 87.0] | 85.2 [71.3 to 101.9]

ADVERSE EVENTS:
Time Frame: Solicited local/general symptoms during the 7-day (Days 0-6) post-vaccination period; AEs during the 30-day (Days 0-29) post-vaccination period; SAEs up to Day 210
Arm/Group | Control Group | GSK692342_F1 Group | GSK692342_F2 Group | GSK692342_F3 Group | GSK692342_F4D1 Group | GSK692342_F4D2 Group
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 2/40 | 0/40 | 2/40 | 0/40
Other Adverse Events (participants affected / at risk) | 10/10 | 9/10 | 40/40 | 39/40 | 39/40 | 38/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control Group (N=10) | GSK692342_F1 Group (N=10) | GSK692342_F2 Group (N=40) | GSK692342_F3 Group (N=40) | GSK692342_F4D1 Group (N=40) | GSK692342_F4D2 Group (N=40)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dengue fever (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Typhoid fever (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Control Group (N=10) | GSK692342_F1 Group (N=10) | GSK692342_F2 Group (N=40) | GSK692342_F3 Group (N=40) | GSK692342_F4D1 Group (N=40) | GSK692342_F4D2 Group (N=40)
Pain (General disorders) | 9 | 5 | 38 | 37 | 37 | 36
Redness (General disorders) | 1 | 2 | 7 | 6 | 6 | 6
Swelling (General disorders) | 1 | 1 | 10 | 10 | 12 | 12
Fatigue (General disorders) | 2 | 1 | 7 | 8 | 13 | 10
Gastro-intestinal symptoms (General disorders) | 3 | 3 | 8 | 9 | 11 | 10
Headache (General disorders) | 5 | 6 | 25 | 27 | 30 | 26
Malaise (General disorders) | 5 | 3 | 23 | 25 | 23 | 26
Myalgia (General disorders) | 3 | 3 | 25 | 23 | 24 | 29
Temperature (Axillary) (General disorders) | 5 | 1 | 17 | 9 | 17 | 28
Nasopharyngitis (Infections and infestations) | 4 | 5 | 15 | 10 | 18 | 16
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 3 | 6 | 13 | 11
Headache (Nervous system disorders) | 2 | 3 | 5 | 7 | 11 | 7
Pyrexia (General disorders) | 1 | 3 | 4 | 4 | 5 | 3
Dizziness (Nervous system disorders) | 2 | 1 | 1 | 5 | 4 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 4 | 1 | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 2 | 2 | 3
Feeling hot (General disorders) | 0 | 0 | 0 | 1 | 4 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 3 | 1 | 1 | 1
Malaise (General disorders) | 0 | 3 | 0 | 0 | 2 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 3 | 1
Toothache (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 3 | 1
Wound (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.